CLINICAL TRIAL: NCT02066142
Title: Tomosynthesis (TS) Versus Ultrasonography (US) in Screening Women With Dense Breast
Brief Title: Tomosynthesis (TS) Versus Ultrasonography (US) in Women With Dense Breast
Acronym: ASTOUND
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Genova (Other)
Collaborators: University of Sydney (Other)
Responsible Party: Principal Investigator, Alberto Tagliafico, Assistant Professor, University of Genova
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PRA20132014
Record Dates: First submitted 2014-02-10; First posted 2014-02-19 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammography; Ultrasonography

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tomosynthesis (Active Comparator): Tomosynthesis will be compared to Ultrasound
  Interventions: Device: 3D mammography (Tomosynthesis)
- Ultrasound (Other): Ultrasound (sensitivity and specificity) will be compared to Tomosynthesis
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: 3D mammography (Tomosynthesis) — Tomosynthesis will be used as normally employed in clinical practice
  Arms: Tomosynthesis
Device: Ultrasound
  Arms: Ultrasound

SUMMARY:
Hypothesis The study aims to demonstrate at least equivalence, or non-significant difference between TS and US in women with dense breast screened negative at 2D Mammography.

If the equivalence between TS and US will be demonstrated, US may be substituted by TS with great benefits for the patients and for the healthcare resources.

Aims

1. Assess if TS may detect additional cancers in dense breast that approximate US detection capability but with less false positive findings than US.
2. If TS detects new cancers in dense breast similarly to US (approximate rate or marginally lower rate), evaluate the the true positive/false positive ratio.
3. Cost-analysis. In case of less false positives detected by TS, the true-positive / false positive trade-off might be strongly in favour of TS with a great potential of costs reduction.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic subjects <50 years of age presenting for mammography, with the exception of those that, on previous mammograms are found to have breast density 1-2 according to the Breast Imaging Reporting and Data System (BIRADS D1-2). - Asymptomatic subjects ≥ 50 years of age who request mammography and have breast density BIRADS 3-4.
* No history of breast cancer - Written informed consent

Exclusion Criteria:

* Pregnant and breast feeding women
* Unable to tolerate breast compression
* Breast implants
* Unable to understand or execute written informed consent
* Unable or unwilling to agree to follow-up during observation period

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2012-12; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
1) Sensitivity of TS | up to 36 months
  We want to verify if TS may detect additional cancers in dense breast that approximate US detection capability but with less false positive findings than US.

SECONDARY OUTCOMES:
2) Specificity of TS | up to 36 months
  If TS detects new cancers in dense breast similarly to US (approximate rate or marginally lower rate), evaluate the the true positive/false positive ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto S Tagliafico, MD, Principal Investigator — UNIGE
Locations (1):
- UNIGE, Genova, Genova, Italy